CLINICAL TRIAL: NCT03478709
Title: Dynamic Arterial Elastance: an Indirect Marker of the Critical Capillary Pressure at the Microcirculatory Level (POEME)
Brief Title: Dynamic Arterial Elastance: an Indirect Marker of the Critical Capillary Pressure at the Microcirculatory Level
Acronym: POEME
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI 2017_843_0012
Record Dates: First submitted 2018-02-28; First posted 2018-03-27 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Arterial Disease
Keywords: vasoplegia; dynamic arterial elastance; microcirculation
MeSH Terms: conditions — Vasoplegia | interventions — Norepinephrine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Volume expansion
  Interventions: Other: volume expansion
- norepinephrine
  Interventions: Other: norepinephrine

INTERVENTIONS:
Other: volume expansion — Volume expansion when the patient has a dependent preload evaluated by a positive leg lever test (variation of more than 10% of the VES). It corresponds to the intravenous administration of 500 ml of Ringer lactate over 10 min.
  Groups: Volume expansion
Other: norepinephrine — Vasopressor agent when the patient has persistent arterial hypotension related to postoperative vasoplegia syndrome. Norepinephrine is administered during persistent hypotension (MAP <60mmHg) despite volume expansion. It corresponds to continuous intravenous norepinephrine administration to obtain a MAP of more than 70 mmHg
  Groups: norepinephrine

SUMMARY:
The measurement of dynamic arterial elastance (Eadyn) was proposed as a marker of vascular tone. It is calculated by the ratio of the respiratory variation of the pulse pressure and the respiratory variation of stroke volume. Despite several clinical studies, no study has really focused on the physiological significance of Eadyn. No study demonstrates at present, if this index is a reflect of macrocirculatory parameters (systemic resistances, blood pressure, arterial elastance, ventricular elastance, ventriculo-arterial coupling) or microcirculatory tone in the capillaries and small arterioles (critical capillary pressure or capillary resistance). the physicians don't know which variables are associated with this index. the hypothesis is that Eadyn is an indirect reflect of capillary pressure (PCC).

DETAILED DESCRIPTION:
The measurement of dynamic arterial elastance (Eadyn) was proposed as a marker of vascular tone. It is calculated by the ratio of the respiratory variation of the pulse pressure and the respiratory variation of stroke volume. Despite several clinical studies, no study has really focused on the physiological significance of Eadyn. No study demonstrates at present, if this index is a reflect of macrocirculatory parameters (systemic resistances, blood pressure, arterial elastance, ventricular elastance, ventriculo-arterial coupling) or microcirculatory tone in the capillaries and small arterioles (critical capillary pressure or capillary resistance). the physicians don't know which variables are associated with this index. One hypothesis is that Eadyn is an indirect reflection of capillary pressure (PCC). The main objective of this project is to study the correlation between the measure of Eadyn and the PCC. The study begins when the physician in charge of the patient decides a hemodynamic treatment (either volume expansion or norepinephrine). The indication of the treatment is left to the discretion of the physician in charge of the patient: volume expansion or vasopressor agent. After verification of inclusion criteria, the physician collects demographic, ventilatory, hemodynamic, cardiac ultrasound data, and the type of treatment initiated (volume expansion, norepinephrine, and their dosages). 15 minutes after the introduction of the therapy and stabilization of the hemodynamic state, a new series of measurements of the aforementioned.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to intensive care, for whom the physician has decided, in accordance with the care protocols of the service, to provide treatment for preload dependence or post-operative vasoplegia syndrome,

  * patients monitored by a central venous catheter, a measurement of blood pressure with continuous monitoring of cardiac output by calibrated analysis of the pulse wave contour (PICCO or EV1000),
  * Patients with sinus heart rate,
  * Patients covered by a social insurance system,
  * Patients who have given their oral consent to participation after complete information

Exclusion Criteria:

* Modification of therapies during the study period,
* Rhythm disorder with PM
* Appearance of cardiac rhythm disturbances (Ac / Fa, Tac / Fa, TV, FV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to intensive care
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-10-22 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
to assess correlation between Eadyn and PCC measure | 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bar S, Nguyen M, Abou-Arab O, Dupont H, Bouhemad B, Guinot PG. Dynamic Arterial Elastance Is Associated With the Vascular Waterfall in Patients Treated With Norepinephrine: An Observational Study. Front Physiol. 2021 May 4;12:583370. doi: 10.3389/fphys.2021.583370. eCollection 2021. PMID 34017263